CLINICAL TRIAL: NCT01478789
Title: Naturalis Clinical Trial for a Novel Phytosterol Formulation
Brief Title: Efficacy of Plant Sterol-Fortified Dairy Product on Plasma Lipid and Plant Sterol Concentrations in Humans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Responsible Party: Principal Investigator, Dr. Peter Jones, Director of the Richardson Centre for Functional Foods and Nutraceuticals, University of Manitoba
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: B2010:096
Record Dates: First submitted 2011-11-17; First posted 2011-11-23 (Estimated); Last update posted 2011-12-21 (Estimated); Status verified 2011-12

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Water dispersible Plant Sterol (WD-PS) (Experimental): WD-PS dairy product (a novel formulation for dispersible free sterols in aqueous media produced)2g/d of free plant sterol
  Interventions: Dietary Supplement: WD-PS intervention phase
- Esterified plant sterol (PS-Ester) (Experimental): PS-Ester enriched dairy product (2g/d free plant sterol)
  Interventions: Dietary Supplement: PS-Ester intervention phase
- placebo (Placebo Comparator): 100 g/d yogurt with no added plant sterol
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: WD-PS intervention phase — 2g/d of free plant sterol in 100g yogurt
  Arms: Water dispersible Plant Sterol (WD-PS)
Dietary Supplement: PS-Ester intervention phase — 2g/d of free plant sterol in 100g yogurt
  Arms: Esterified plant sterol (PS-Ester)
Dietary Supplement: placebo — 100g/d yogurt with no added plant sterol
  Arms: placebo

SUMMARY:
The aim of this clinical study was to determine the efficacy on plasma cholesterol-lowering of a water dispersible formulation of plant sterol (WD-PS) preparation versus plant sterol esters (PS-ester), consumed within dairy products.

DETAILED DESCRIPTION:
Forty-seven hyperlipidemic subjects (25 males and 22 females, age 19-75 years at baseline) completed the double-blind, randomized, crossover study.

ELIGIBILITY:
Inclusion Criteria:

* healthy individuals aged 19-60 yr
* plasma LDL-C levels > 3.0mmol/l
* TG < 4.5mmol/l
* body mass index (BMI) between 20 and 30 kg/m2.

Exclusion Criteria:

* history of recent or chronic use of oral hypolipidemic therapy, including fish oils, or probucol within the last 3 months
* history of chronic use of alcohol (>2 drinks/d)
* smoking
* myocardial infarction, coronary artery bypass, sitosterolaemia, kidney disease, liver disease or other major surgical procedures within the last six months

Ages: 19 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2010-09; Primary Completion 2011-02 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Lipid Profile | Change from Baseline in lipid profile at 4 weeks (end of the phase)

CONTACTS AND LOCATIONS:
Locations (1):
- Richarson Centre for Funtional Foods and Nutraceuticals, Winnipeg, Manitoba, Canada